CLINICAL TRIAL: NCT05660434
Title: Using Aromatherapy for Comfort, Ease, and Stress for Adults Being Treated for Substance Use Disorder in North Central Appalachia: A Randomized Controlled Trial
Brief Title: Using Aromatherapy in Substance Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: West Virginia Nurses Association (Other)
Responsible Party: Principal Investigator, Marian Reven, Assistant Professor, Principle Investigator, West Virginia University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2204562633
Record Dates: First submitted 2022-11-18; First posted 2022-12-21 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Substance Use Disorders
Keywords: social and behavioral; randomized; questionnaires; aroma therapy
MeSH Terms: conditions — Substance-Related Disorders; Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The person enrolling is masked to the assignment. No need to mask for aroma inhaler as participants receive materials through the mail and do not interact with other participants. No sham inhaler is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Adults (>18 years) who are currently receiving treatment for substance use disorder (SUD) in the outpatient treatment program at West Virginia University Chestnut Ridge Center (WVUCRC) (n = 340 approx.). In addition, participants can be at any level of treatment, including peer recovery coach program. Inclusion criteria are patients diagnosed with SUD who have completed intensive acute phase 1 treatment, and who desire to pursue continuous recovery phases (per facility protocol). All participants must be alert and oriented, provide written consent, and be able to read and write English. Exclusion criteria are patients diagnosed with severe mental illness (who cannot consent to participate), have a medical history of asthma or other serious respiratory disease, and known allergy to citrus.
  Interventions: Other: Aroma Inhaler with Bergamot essential oil
- Control Group (No Intervention): Adults (>18 years) who are currently receiving treatment for SUD in the outpatient treatment program at West Virginia University Chestnut Ridge Center (WVUCRC) (n = 340 approx.). In addition, participants can be at any level of treatment, including peer recovery coach program. Inclusion criteria are patients diagnosed with SUD who have completed intensive acute phase 1 treatment, and who desire to pursue continuous recovery phases (per facility protocol). All participants must be alert and oriented, provide written consent, and be able to read and write English. Exclusion criteria are patients diagnosed with severe mental illness (who cannot consent to participate), have a medical history of asthma or other serious respiratory disease, and known allergy to citrus.

INTERVENTIONS:
Other: Aroma Inhaler with Bergamot essential oil — The intervention group will receive an aroma inhaler and logbook to use three times a day for 7 days and complete pre and post surveys for comfort, ease, and stress.
  Arms: Intervention Group

SUMMARY:
The purpose of this clinical trial study is to see if Bergamot, an aroma therapy essential oil, has any effect on comfort, ease, and stress. Participants will be asked to use a bergamot aroma inhaler, which is a small tube about the size of a lipstick container, at least three times a day for one week. Comfort, ease, and stress will be measured with self-report survey at the beginning and at the end of the week. In addition, participants will be asked to complete a daily logbook to record use of the inhaler. The study lasts for one week (7 days). The aims of this study are to explore the effects of Bergamot essential oil on comfort, ease, and stress in adults in a substance use disorder (SUD) treatment program, and to evaluate the feasibility of this type of aroma therapy intervention.

DETAILED DESCRIPTION:
Statement of purpose: The purpose of the study is to examine the effect of an aromatic intervention using bergamot essential oil on comfort, ease, and stress in adults in a SUD recovery program

Research Question: What are differences in comfort, ease, and stress for persons in a substance use disorder program who receive aromatic intervention and for those who do not?

Conceptual framework: An integrated theoretical framework combining the theory of comfort (Kolcaba, 2003) and the concept of welcoming ease (Reven, 2022) will be used as theoretical guidance for this study.

Aims and Objectives: Specific Aim #1: Evaluate the feasibility and acceptability of an aromatherapy intervention by examining recruitment, enrollment and retention rates, intervention fidelity, and cost analysis. Specific Aim #2: Pilot test bergamot essential oil intervention with adults in a substance use disorder recovery program.

Background: Appalachia is at the epicenter of the opioid addiction crisis with hardly a family left untouched by the devastating consequences. Those who make it to recovery programs are often plagued by anxiety and depression. Those in treatment have identified increasing the level of comfort during substance use recovery as vital. Integrating aromatherapy could help improve perception of comfort and reduce stress thus enhancing recovery program progression.

Methods: The study uses a parallel-randomized control group comparison design. Data will be collected from participants daily and post intervention. For Aim #1, descriptive and bivariate analysis will be conducted. Statistical assumptions will be tested. Sample demographics will be reported. For Aim #2, descriptive statistics will be used as well as participant recruitment, enrollment, and retention rates. Reasons for non-participation and attrition will be recorded. Percentage of intervention consistency will be calculated and cost of the intervention will be determined.

Timeline: The proposed study would begin as soon as grant funding is available with projected timeline being August 2022 to December 2023.

ELIGIBILITY:
Inclusion Criteria:

* Participants can be at any level of treatment, including peer recovery coach program at West Virginia University Comprehensive Opioid Addiction Treatment (COAT) program
* All participants must be alert and oriented
* Provide written consent
* Able to read and write English

Exclusion Criteria:

* Have a medical history of asthma or other serious respiratory disease
* Known allergy to citrus.
* Dislike of Bergamot

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marian Reven, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be maintained by the primary investigator, and will be analyzed and reported by this individual only.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 45 | 55
Completed | 43 | 54
Not Completed | 2 | 1
Not completed — Never obtained study materials | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Adults (>18 years) who are currently receiving treatment for SUD in the outpatient treatment program at West Virginia University Chestnut Ridge Center (WVUCRC) (n = 340 approx.). In addition, participants can be at any level of treatment, including peer recovery coach program. Inclusion criteria are patients diagnosed with SUD who have completed intensive acute phase 1 treatment, and who desire to pursue continuous recovery phases (per facility protocol). All participants must be alert and oriented, provide written consent, and be able to read and write English. Exclusion criteria are patients diagnosed with severe mental illness (who cannot consent to participate), have a medical history of asthma or other serious respiratory disease, and known allergy to citrus.
  Aroma Inhaler with Bergamot essential oil: The intervention group will receive an aroma inhaler and logbook to use three times a day for 7 days and complete pre and post surveys for comfort, ease, and stress.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 45 | 55 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 55 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 35 | 61
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 44 | 52 | 96
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Examine Feasibility (Eligible Participant Recruitment)
Description: Determine feasibility by assessing the number of eligible participants recruited.
Time Frame: Up to 18 months
Population: The numbers above reflect all patients that were deemed eligible per criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 45 | 55
Participants | 45 | 55

2. Primary Outcome: Examine Feasibility (Eligible Participant Enrollment)
Description: Determine feasibility by assessing how many eligible participants enroll.
Time Frame: Up to 18 months
Population: The numbers above reflect all patients that were deemed eligible per criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 45 | 55
Participants | 45 | 55

3. Primary Outcome: Examine Feasibility (Participant Retention)
Description: Determine feasibility by assessing count of participants retained.
Time Frame: Up to 18 months
Population: 3 participants never obtained study materials
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 45 | 55
Participants | 43 | 54

4. Primary Outcome: Examine Fidelity of the Intervention
Description: Determine fidelity by assessing the count of participants that completed the intervention as directed as shown in the daily logbook.
Time Frame: Up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 45 | 55
Participants | 45 | 55

5. Secondary Outcome: Change in Perceived Comfort Level
Description: The concept of comfort is operationalized by the Generalized Comfort Questionnaire (GCQ). This incorporates a Likert scale from 1 to 6 with 1 being the least agreement with the statement and 6 being the most agreement with the statement. The investigators are looking at a change in comfort from before the intervention to after the intervention. There were 28 questions in this scale with a total score between 28 and 168. There are 3 subscales of Relief (8 questions) , Ease (10 questions), and Transcendence (10 questions). A higher score post test cumulative or as subscales indicates more agreement with the statements of overall comfort and its subscales.
Time Frame: Pre test prior to day 1 to Post test after 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 45 | 55
score on a scale
  Before Intervention | 116.29 (21.798) | 114.17 (22.050)
  After Intervention | 117.91 (20.599) | 114.84 (21.683)

6. Secondary Outcome: Change in Perceived Ease Level
Description: The concept of ease is measured using the Ease measure. This is assessed using a Likert scale from 1 to 4. There is only one score reported for this measure, no subscales. The investigators are looking at a change in ease from before the intervention to after the intervention. There are 20 questions with a range of scores between 20 and 80. The lower score indicates less agreement with the statement about ease. A higher score indicates more agreement. A higher score post test indicates an improvement.
Time Frame: Pre test prior to day 1 to Post test after 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 45 | 55
score on a scale
  Before Intervention | 53.04 (9.925) | 53.88 (8.993)
  After Intervention | 57.21 (11.482) | 55.58 (8.212)

7. Secondary Outcome: Change in the Depression, Anxiety, and Stress Scale (DASS-21)
Description: The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items. This is assessed using a Likert scale from 0 to 3 with 0 being the least amount of stress and 3 being the highest amount of stress. Scores range from 0 to 63 with lower score indicating less agreement with statements and 63 indicating higher score in agreement with statements. A lower score indicates improvement in DASS.
Time Frame: Pre test prior to day 1 to Post test after 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 45 | 55
score on a scale
  Before Intervention | 20.49 (11.482) | 20.28 (10.747)
  After Intervention | 18.54 (10.404) | 21.34 (10.953)

8. Secondary Outcome: Visual Analogue Scale to Assess Daily Perceived Comfort
Description: The Visual Analogue Scale (VAS) is used as a daily measure of comfort. It provides validation for the GCQ using a 100mm line where Comfort is rated using a mark on the line between 0 and 100 "I feel as comfortable as possible" with 0 being the least comfortable and 100 being the most comfortable.
Time Frame: 7 days
Population: Per Protocol only 25 participants were included in the Intervention group for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 25 | 42
score on a scale
  Day 1 | 66.72 (18.729) | 49.02 (26.386)
  Day 7 | 80.68 (11.707) | 55.71 (26.516)

ADVERSE EVENTS:
Time Frame: 7 Days
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/55
Other Adverse Events (participants affected / at risk) | 0/45 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT05660434/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT05660434/ICF_001.pdf